CLINICAL TRIAL: NCT00731198
Title: Drotaverine Hydrochloride Versus Hyoscine-N-butylbromide for Duodenal Antimotility During ERCP: a Prospective, Multicenter Randomized Controlled Trial
Brief Title: Drotaverine Hydrochloride Versus Hyoscine-N-butylbromide for Duodenal Antimotility During Endoscopic Retrograde Cholangiopancreatography (ERCP)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Zhaoshen Li, Changhai Hospital, Second Military Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Changhai-080615
Record Dates: First submitted 2008-08-06; First posted 2008-08-08 (Estimated); Results first posted 2009-12-23 (Estimated); Last update posted 2010-09-08 (Estimated); Status verified 2009-11

CONDITIONS: ERCP; Pancreatic Diseases; Bile Duct Diseases
Keywords: ERCP; Drotaverine hydrochloride; Hyoscine-N-butylbromide
MeSH Terms: conditions — Pancreatic Diseases; Bile Duct Diseases | interventions — drotaverin; Butylscopolammonium Bromide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Drotaverine hydrochloride
  Interventions: Drug: Drotaverine hydrochloride
- 2 (Active Comparator): Hyoscine-N-butylbromide
  Interventions: Drug: Hyoscine-N-butylbromide

INTERVENTIONS:
Drug: Drotaverine hydrochloride — Drotaverine hydrochloride 40mg was administered intravenously 15 minutes before ERCP
  Other Names: No-spa
  Arms: 1
Drug: Hyoscine-N-butylbromide — Hyoscine-N-butylbromide 20mg was administered intravenously 15 minutes before ERCP.
  Other Names: Scopolamine Butylbromide
  Arms: 2

SUMMARY:
The aim of the present study was to evaluate the use of drotaverine hydrochloride versus hyoscine-N-butylbromide in reducing duodenal motility during diagnostic and therapeutic ERCP.

DETAILED DESCRIPTION:
ERCP is an important endoscopic technique in the diagnosis and treatment of pancreatic and biliary diseases. Duodenal peristalsis can make cannulation of the papilla and the necessary therapeutic procedures difficult. Intravenous hyoscine-N-butylbromide is often used during ERCP to inhibit duodenal motility and enhance cannulation in China. However, the pharmaceutical agent is occasionally associated with serious complications such as cardiovascular events or anaphylactic shock. Hyoscine-N-butylbromide may also affect the ocular, urinary, and salivary systems.

Drotaverine hydrochloride is an analogue of papaverine with smooth muscle relaxant properties. It is a non-anticholinergic antispasmodic, which selectively inhibits phosphodiesterase IV and is accompanied by a mild calcium channel-blocking effect. Adverse effects with drotaverine hydrochloride, such as hypotension, vertigo, nausea, and palpitation, are mostly mild. It can be supposed that intravenous drotaverine hydrochloride might be a feasible antimotility alternative to intravenous hyoscine-N-butylbromide in ERCP. But there is no clear evidence to recommend the use of drotaverine hydrochloride as an antispasmodic during ERCP.

The aim of the present study was to evaluate the use of drotaverine hydrochloride versus hyoscine-N-butylbromide in reducing duodenal motility during diagnostic and therapeutic ERCP. The effects of drotaverine hydrochloride on facilitative cannulation and its adverse effects were also compared to hyoscine-N-butylbromide.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing ERCP above the age of 18 years

Exclusion Criteria:

* Patient with Billroth II gastrectomy
* Known previous sphincterotomy
* Active acute pancreatitis before ERCP
* Ongoing acute cholangitis before ERCP
* Hypotension (systolic blood pressure < 100 mmHg)
* Second-degree and third-degree atrioventricular block
* Heart failure
* Glaucoma
* Obstructive uropathy
* Impaired renal function (serum creatinine > 133μmol/L)
* Pregnant or breastfeeding women

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 650 (Actual)
Dates: Start 2008-08; Primary Completion 2009-03 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoshen Li, MD, Principal Investigator — Changhai Hospital
Locations (4):
- China (4):
  - Fujian Provincial Hospital, Fuzhou
  - The First People's Hospital of Hangzhou, Hangzhou
  - Heilongjiang Provincial Hospital, Harbin
  - Changhai Hospital, Second Military Medical University, Shanghai

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: Drotaverine hydrochloride
- Active Comparator: Hyoscine-N-butylbromide
Period: Overall Study
Arm/Group | Experimental | Active Comparator
Started | 325 | 325
Completed | 319 | 319
Not Completed | 6 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental | Active Comparator | Total
Number analyzed (Participants) | 325 | 325 | 650
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 205 | 197 | 402
  >=65 years | 120 | 128 | 248
Age Continuous [Mean (Standard Deviation); unit: years] | 56.98 (15.75) | 59.20 (16.14) | 58.09 (15.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 139 | 173 | 312
  Male | 186 | 152 | 338
Region of Enrollment [Number; unit: participants]
  China | 325 | 325 | 650

OUTCOME MEASURES:

1. Primary Outcome: The Grades of the Number of Duodenal Contractions
Description: a duodenal motility grade was determined as follows: 0 = no motility; 1 = less than five contractions/minute; 2 = 5 to 10/minute; 3 = 11 to 15/minute; 4 = continuous.
Time Frame: Intra-procedure
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Experimental | Active Comparator
Number analyzed (Participants) | 319 | 319
scores on a scale | 1.13 (0.89) | 1.17 (0.82)

2. Secondary Outcome: Cannulation Time
Time Frame: Intra-procedure
Reporting Status: Not Posted

3. Secondary Outcome: Percentage of Successful Selective Cannulation
Time Frame: Intra-procedure
Reporting Status: Not Posted

4. Secondary Outcome: Frequency of Post-ERCP Complications
Time Frame: 48 hours after ERCP
Reporting Status: Not Posted

5. Secondary Outcome: Side Effects
Time Frame: Intra-procedure and 24 hours after ERCP
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Experimental | Active Comparator
Serious Adverse Events (participants affected / at risk) | 0/319 | 0/319
Other Adverse Events (participants affected / at risk) | 0/319 | 0/319

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No